CLINICAL TRIAL: NCT06561854
Title: Free Regimen of Dexamethasone as Initial Therapy for Advanced Relapsed/Refractory Multiple Myeloma: an Open-label Randomized, Non-inferiority, Controlled Trial
Brief Title: Study Comparing Therapy for Advanced Relapsed/Refractory Multiple Myeloma With and Without Dexamethasone
Acronym: FREEDOM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP231089; 2024-510981-18-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-07; First posted 2024-08-20 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Multiple Myeloma; Relapse Multiple Myeloma
Keywords: Multiple myeloma; Relapse; Dexamethasone; Isatuximab; Pomalidomide; Carfilzomib
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone-free (Experimental): Dexamethasone will be stopped after the first 2 cycles (in both ICARIA and IKEMA schemas).
  ICARIA shemas :
  dexamethasone isatuximab pomalidomide
  IKEMA shemas :
  dexamethasone isatuximab carfilzomib
  Interventions: Drug: Dexamethasone
- Dexamethasone (No Intervention): Dexamethasone will not be discontinued (in both ICARIA and IKEMA shemas).
  ICARIA schema :
  dexamethasone isatuximab pomalidomide
  IKEMA schema :
  dexamethasone isatuximab carfilzomib

INTERVENTIONS:
Drug: Dexamethasone — ICARIA schema :
  40mg (20mg for ≥75yr) on day 1, 8, 15, 22 of each cycle plus
  IKEMA schema :
  20 mg on day 1-2, day 8-9, day 15-16 and day 22-23 of each cycle
  For subjects older than 75 years or underweight (BMI <18.5), the dexamethasone dose may be administered at a total dose of 20 mg weekly.
  In both schema (ICARIA or IKEMA), dexamethasone will be administrated up to 2 cycle (Arm 1) or until disease progression (Arm2)
  Other Names: Neofordex
  Arms: Dexamethasone-free

SUMMARY:
Patients with relapsed/refractory symptomatic multiple myeloma who meet all inclusion criteria, will be randomized 1:1 to receive either standard of care chemotherapy (IKEMA or ICARIA) and dexamethasone until disease progression ("dexamethasone arm", arm A) or standard of care chemotherapy (IKEMA or ICARIA) and dexamethasone with dexamethasone discontinuation from the 3rd cycle of treatment (after 8 weeks) ("dexamethasone-free arm", arm B).

In most centers, IKEMA and ICARIA schema can be adapted according to the standard of care in each center Choice between the ICARIA and IKEMA schema is at the discretion of the investigator, in compliance with each drug's SmPC, but must be performed before randomisation for the purpose of stratification.

DETAILED DESCRIPTION:
Patients with relapsed/refractory symptomatic multiple myeloma who meet all inclusion criteria, will be randomized 1:1 to receive either standard of care chemotherapy (IKEMA or ICARIA) and dexamethasone until disease progression ("dexamethasone arm", arm A) or standard of care chemotherapy (IKEMA or ICARIA) and dexamethasone with dexamethasone discontinuation from the 3rd cycle of treatment (after 8 weeks) ("dexamethasone-free arm", arm B).

In most centers, IKEMA and ICARIA schema are as follow, but can be adapted according to the standard of care in each center Choice between the ICARIA and IKEMA schema is at the discretion of the investigator, in compliance with each drug's SmPC, but must be performed before randomisation for the purpose of stratification.

1. ICARIA schema:

   * dexamethasone: 40mg (20mg for ≥75yr) on day 1, 8, 15, 22 of each cycle plus
   * isatuximab: 10mg/kg on day 1, 8, 15, 22 in C1 subsequently on day 1, 15; plus
   * pomalidomide: 4mg on days 1-21 of 28-day cycle.
2. IKEMA schema:

   * dexamethasone: 20 mg on day 1-2, day 8-9, day 15-16 and day 22-23 of each cycle;
   * isatuximab: 10 mg/kg on day 1, 8, 15, 22 in C1, then Q2W;
   * carfilzomib: 20 mg/m² on day 1-2; 56 mg/m² day 8-9, day, 15-16 in C1; 56 mg/m² on day 1-2, day 8-9, day 15-16 all subsequent cycles.

In the dexamethasone arm (standard of care):

Dexamethasone: will be given on each cycle

In the dexamethasone-free arm (experimental arm):

Dexamethasone: will be only given on cycle 1 and cycle 2 Supportive care: will be administered according to each participating center's usual practice, in both arms The aim of the current protocol is to investigate whether administration of dexamethasone for a very limited period (2 cycles) combined with standard treatment for relapsed/refractory MM is not inferior to the continuous administration of the combination until disease progression. In this study some patients may have a similar OS while receiving a shorter duration of dexamethasone treatment. This study may allow delivery of a shorter duration of dexamethasone for the treatment of relapsed MM.

The foreseeable risks are those of an earlier relapse in patients receiving a short duration of dexamethasone (8 weeks) compared to the situation where they would have received the dexamethasone until disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years old)
2. Documented MM in relapse according to standard criteria.
3. All patients must have received between 1 to 3 prior therapies for MM (a prior therapy is defined as 2 or more cycles of therapy given as a MM treatment plan)

   * Eligible for one of the following antibody-based approved combinations:

     1. ICARIA schema: isatuximab, pomalidomide and dexamethasone.
     2. IKEMA schema: isatuximab, carfilzomib and dexamethasone
4. Subject must have achieved a response (PR or better) to the prior regimen.
5. ECOG Performance Status score of 0, 1, or 2.
6. For subjects experiencing toxicities resulting from previous therapy (including peripheral neuropathy), the toxicities must have been resolved or stabilized.
7. Signed informed consent

Exclusion Criteria:

1. Contraindications to investigational medicinal products or auxiliary medicinal product
2. Evidence of refractoriness or intolerance to anti-CD38 monoclonal antibodies.
3. Previous treatment according to the ICARIA schema with pomalidomide or IKEMA schema with carfilzomib
4. Allogenic hematopoietic cell transplant (HCT, regardless of timing).
5. Planned to undergo an hematopoietic cell transplant prior to progression of disease ie, these patients should not be enrolled in order to reduce disease burden prior to transplant.
6. History of malignancy (other than MM) within 3 years before the date of randomization (exceptions are squamous and basal cell carcinomas of the skin, carcinoma in situ of the cervix, or malignancy that in the opinion of the Investigator is considered cured with minimal risk of recurrence within 3 years).
7. Known MM meningeal Involvement.
8. Plasma cell leukemia (>2.0 × 109/L circulating plasma cells by standard differential) or Waldenström's macroglobulinemia or POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes) or amyloidosis.
9. Any concurrent medical condition or disease (e.g., active systemic infection) that is likely to interfere with study procedures or results, or that, in the opinion, of the Investigator would constitute a hazard by participating in this study.
10. Uncontrolled chronic obstructive pulmonary disease (COPD)
11. Clinically significant cardiac disease.
12. Seropositive for hepatitis B with positive PCR
13. Seropositive for human immunodeficiency virus (HIV) or hepatitis C
14. Lactation
15. Participation to another interventional clinical trial
16. Inability to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
overall response rate (ORR). | At the end of Cycle 6 of salvage therapy (each cycle is 28 days)
  Response rate will be evaluated according to the IMWG criteria, after six 28 days cycles of salvage therapy.

SECONDARY OUTCOMES:
best overall response rate (ORR) | 2 years
  Response rate will be evaluated according to the IMWG criteria, during or after the study treatment at the time of data cutoff. Patients will be followed every 4 weeks (with either a medical visit or only an outpatient blood test) until disease progression and then every 12 weeks until final 2 years.
Time To Progress (TTP) | 2 years
  Time To Progress defined as the duration from the date of randomization to progressive disease, according to the IMWG criteria
Progression free survival (PFS) | 2 years
  Progression free survival is defined as the duration from the date of randomization to either progressive disease, according to the IMWG critera or death, at 2 years after randomization.
Overall survival OS | 2 years
  which is defined as the time between randomization and death due to any cause. Patients, who die, regardless of the cause of death, will be considered to have had an event even if they were lost to follow-up for an extended time
Quality of Life (QoL) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad MOHTY, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service d'hématologie clinique et thérapie cellulaire, Saint-Antoine Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided